CLINICAL TRIAL: NCT01532739
Title: Neuropsychological Intervention for a Seniors Mental Health Population With Mild Cognitive Impairment
Brief Title: Making Memory Better for Seniors With Mild Cognitive Impairment
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: Nova Scotia Health Research Foundation (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CDHA-RS/2012-227
Record Dates: First submitted 2012-02-10; First posted 2012-02-14 (Estimated); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Mild Cognitive Impairment
Keywords: Mild Cognitive Impairment; Aging; Memory; Executive Function; Cognitive Intervention; Memory Training; Mental Health
MeSH Terms: conditions — Cognitive Dysfunction; Psychological Well-Being | interventions — Cognitive Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive training (Experimental)
  Interventions: Behavioral: Cognitive training
- No cognitive training (No Intervention)

INTERVENTIONS:
Behavioral: Cognitive training — The cognitive training consists of 10 weekly 2-hour sessions. It is run with groups of MCI participants and their study partners (who help with reinforcing the strategies in everyday activities). The program provides information about memory and lifestyle factors in the first two weeks, followed by training and practice over the next eight weeks on empirically-supported cognitive strategies known to be effective at supporting day-to-day remembering in MCI. Participants learn to apply a core set of strategies (spaced retrieval, memory book logging) across a variety of common memory problems (e.g., remembering names, appointments, etc). To enhance the likelihood that these strategies will transfer to other settings beyond training, participants are also taught a memory problem solving approach that will cue them to recognize situations in which they need to: (1) stop and remember something, (2) select and apply an appropriate memory strategy, and (3) monitor that it is working.
  Arms: Cognitive training

SUMMARY:
The purpose of this study is to investigate the feasibility and effectiveness of a cognitive training group in individuals with Mild Cognitive Impairment, using a new paradigm that will optimize ecological validity by (1) focusing on everyday memory problems, (2) supplementing traditional memory training with the teaching of an empirically-supported problem-solving approach, and (3) employing a clinically representative sample of individuals with MCI (e.g., not excluding those with mild affective symptoms).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Mild Cognitive Impairment

Exclusion Criteria:

* Clinical diagnosis of dementia
* History of neurological conditions known to impair cognition
* History of alcohol or drug abuse
* History of chronic psychiatric illness
* Current symptoms of moderate to severe depression (Geriatric Depression Scale >19) or anxiety (Beck Anxiety Inventory >15)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-12-05 (Actual); Primary Completion 2025-12-05 (Estimated); Study Completion 2025-12-05 (Estimated)

PRIMARY OUTCOMES:
Change in everyday memory functioning | Measured at baseline and months 3, 5, 8
  Rivermead Behavioural Memory Test (3rd Edition)

SECONDARY OUTCOMES:
Change on traditional memory testing | Measured at baseline and months 3, 5, 8
  California Verbal Learning Test (2nd Edition)
Change in memory perception | Measured at baseline and months 3, 5, 8
  Multifactorial Metamemory Questionnaire
Change in mood (i.e., self-report symptoms of depression) | Measured at baseline and months 3, 5, 8
  Geriatric Depression Scale
Change in mood (i.e., self-report symptoms of anxiety) | Measured at baseline and months 3, 5, 8
  Beck Anxiety Inventory
Change in other psychiatric symptoms (informant-report) | Measured at baseline and months 3, 5, 8
  Neuropsychiatric Inventory
Change in quality of life | Measured at baseline and months 3, 5, 8
  Zarit Burden Interview
Change in caregiver burden | Measured at baseline and months 3, 5, 8
  Zarit Burden Interview
Feasibility | Measured at end of study
  Recruitment, retention, and compliance rates

CONTACTS AND LOCATIONS:
Overall Officials: Karen A Chipman, PhD, Principal Investigator — Nova Scotia Health Authority
Locations (1):
- Neuropsychology Service, Nova Scotia Hospital, Dartmouth, Nova Scotia, Canada